CLINICAL TRIAL: NCT00329173
Title: A 6-Week Open-Label, Randomised, Multicentre, Phase IIIb, Parallel-Group Study to Compare the Efficacy and Safety of Rosuvastatin (10 mg) With Atorvastatin (20 mg) in Subjects With Hypercholesterolaemia and Either a History of CHD or Clinical Evidence of CHD
Brief Title: PULSAR - A Prospective Study to Evaluate the Utility of Low Doses of the Statins Atorvastatin and Rosuvastatin.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4522IL/0102; PULSAR; D3569C00001
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium; Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin
Drug: Atorvastatin

SUMMARY:
To compare reduction of LDL-C and safety between 10mg rosuvastatin and 20mg atorvastatin after 6 weeks treatment

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 or over.
* A history of CHD or clinical evidence of atherosclerosis (diabetic or non-diabetic) or a CHD risk equivalent (10-year risk score > 20% for CHD as described in NCEP ATP III guidelines1.

Exclusion Criteria:

* History of statin induced myopathy, or serious hypersensitivity reaction to other HMG-CoA reductase inhibitors (statins), including rosuvastatin
* Pregnancy
* History of homozygous familial hypercholesterolaemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2003-11; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Reduction in LDL-c after 6 weeks

SECONDARY OUTCOMES:
Changes in other lipids and lipoproteins
Achievement of NCEP -ATP III target goal LDL-Cholesterol and non HDL-C
Achievement of EAS LDL-c and non HDL-C target goals after 6 weeks treatment.
Comparison of cost effectiveness and also safety

CONTACTS AND LOCATIONS:
Overall Officials: Crestor Medical Science Director, MD, Study Director — AstraZeneca